CLINICAL TRIAL: NCT00113087
Title: Trial of ACE Inhibition in Infants With Single Ventricle (A Trial Conducted by the Pediatric Heart Network)
Brief Title: Trial of Angiotensin Converting Enzyme Inhibition in Infants With Single Ventricle--Pediatric Heart Network
Acronym: ISV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Pediatric Heart Network (Other)
Responsible Party: Lynn Sleeper, PI, New England Research Institutes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 177; U01HL068270 (NIH); U01HL068279 (NIH); U01HL068281 (NIH); U01HL068285 (NIH); U01HL068288 (NIH); U01HL068290 (NIH); U01HL068292 (NIH); U01HL068269 (NIH)
Record Dates: First submitted 2005-06-03; First posted 2005-06-06 (Estimated); Results first posted 2010-09-16 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Heart Defects, Congenital; Heart Failure, Congestive
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure | interventions — Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enalapril (Active Comparator): Enalapril (angiotensin converting enzyme inhibitor)
  Interventions: Drug: Enalapril
- Placebo (Placebo Comparator): Placebo (Ora-Plus and Ora-Sweet)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enalapril — Enalapril to target dose of .4mg/kg/day divided to twice per day (BID)
  Arms: Enalapril
Drug: Placebo — Participants will receive placebo
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of administering an angiotensin converting enzyme inhibitor (ACE-I) (enalapril) to infants with a functional single ventricle. The study will also compare the effect of ACE-I therapy to placebo on somatic growth and compare the effect of ACE-I therapy to placebo on signs and symptoms of heart failure, neurodevelopmental and functional status, ventricular geometry, function, and atrioventricular (AV) valve regurgitation. In addition, the study will determine the relationship between genetic polymorphisms linked to ventricular hypertrophy (enlarged heart) and the response to ACE-I therapy and compare the incidence of adverse events in subjects treated with ACE-I with those in subjects treated with placebo.

DETAILED DESCRIPTION:
BACKGROUND:

Growth impairment is common in infants and children with congenital heart disease, most often in the presence of congestive heart failure and/or cyanosis. Growth failure is noted in many infants with a single ventricle who manifest both cyanosis and heart failure that commonly persist after palliative surgery. Whether this impairment is related to persistent or progressive abnormalities in cardiac structure and function is not known. ACE-Is are widely used in the treatment of infants with severe congestive heart failure to improve cardiac function and somatic growth. The ability of an ACE-I to improve somatic growth in infants with a single ventricle has not been previously studied.

This study has been approved by the Institutional Review Boards/Research Ethics Boards of all participating clinical centers:

Hospital for Sick Children, Toronto, Canada

Children's Hospital Boston, Boston, MA

Columbia College of Physicians and Surgeons, New York, NY

Children's Hospital of Philadelphia, Philadelphia, PA

Duke University Medical Center, Durham, NC

Brody School of Medicine at East Carolina University, Greenville, NC

Wake Forest Baptist Medical Center, Winston Salem, NC

Medical University of South Carolina, Charleston, SC

Primary Children's Medical Center, Salt Lake City, UT

Children's Hospital of Wisconsin, Milwaukee, WI

Cincinnati Children's Hospital Medical Center, Cincinnati, OH

DESIGN NARRATIVE:

This is a prospective, randomized, double-blind, placebo-controlled trial of ACE-I in infants with a single ventricle. After stratification by ventricular anatomy, neonates will be randomly assigned to receive enalapril or placebo and then followed for 14 months.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 45 days of age
* Age greater than 1 week if born at 35 weeks gestation
* Single ventricle physiology
* Stable systemic and pulmonary blood flow
* Planned Glenn shunt surgery (or variant known as hemi-Fontan)

Exclusion Criteria:

* Birth weight less than or equal to 2.5 kg if gestational age is greater than or equal to 38 weeks
* Birth weight less than the 10th percentile for gestational age if gestational age is 35 to 37 weeks
* Less than 35 weeks gestation
* Anatomic diagnosis of pulmonary atresia with intact ventricular septum
* Less than 3 days after palliative cardiac surgical procedure, if performed
* Aortic oxygen saturation less than 65%
* Current mechanical ventilatory support
* Current intravenous inotropic support
* Creatinine greater than 1.0 mg/dL
* Absolute neutrophil count less than 1,000 cells/mL
* Chromosomal or recognizable phenotypic syndrome of noncardiac congenital abnormalities associated with growth failure (e.g., Trisomy 21, Noonan's syndrome, Turner's syndrome)
* Prior ACE inhibitor use for greater than 7 consecutive days

Max Age: 45 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2003-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Page Anderson, MD, Principal Investigator — Duke University Medical Center, Durham, NC; Daphne Hsu, MD, Principal Investigator — The Children's Hospital at Montefiore, NYC, NY; Brian McCrindle, MD, Principal Investigator — The Hospital for Sick Children; LuAnn Minich, MD, Principal Investigator — Primary Children's Hospital, Salt Lake City, UT; Jane Newburger, MD, Principal Investigator — Children's Hospital Boston, Boston, MA; J. Philip Saul, MD, Principal Investigator — Medical University of South Carolina; Lynn Sleeper, Sc.D., Principal Investigator — New England Research Institute, Watertown, MA; Victoria Vetter, MD, Principal Investigator — Children's Hospital of Philadelphia, Philadelphia, PA; Woodrow Benson, MD, Principal Investigator — Cincinnati Children's Medical Center, Cincinnati, OH
Locations (9):
- United States (8):
  - Children's Hospital Boston, Boston, Massachusetts
  - Columbia College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Miller TA, Zak V, Shrader P, Ravishankar C, Pemberton VL, Newburger JW, Shillingford AJ, Dagincourt N, Cnota JF, Lambert LM, Sananes R, Richmond ME, Hsu DT, Miller SG, Zyblewski SC, Williams RV; Pediatric Heart Network Investigators. Growth Asymmetry, Head Circumference, and Neurodevelopmental Outcomes in Infants with Single Ventricles. J Pediatr. 2016 Jan;168:220-225.e1. doi: 10.1016/j.jpeds.2015.09.041. Epub 2015 Oct 17. PMID 26490132
- [Derived] Ravishankar C, Zak V, Williams IA, Bellinger DC, Gaynor JW, Ghanayem NS, Krawczeski CD, Licht DJ, Mahony L, Newburger JW, Pemberton VL, Williams RV, Sananes R, Cook AL, Atz T, Khaikin S, Hsu DT; Pediatric Heart Network Investigators. Association of impaired linear growth and worse neurodevelopmental outcome in infants with single ventricle physiology: a report from the pediatric heart network infant single ventricle trial. J Pediatr. 2013 Feb;162(2):250-6.e2. doi: 10.1016/j.jpeds.2012.07.048. Epub 2012 Aug 30. PMID 22939929
- [Derived] Cnota JF, Allen KR, Colan S, Covitz W, Graham EM, Hehir DA, Levine JC, Margossian R, McCrindle BW, Minich LL, Natarajan S, Richmond ME, Hsu DT; Pediatric Heart Network Investigators. Superior cavopulmonary anastomosis timing and outcomes in infants with single ventricle. J Thorac Cardiovasc Surg. 2013 May;145(5):1288-96. doi: 10.1016/j.jtcvs.2012.07.069. Epub 2012 Aug 28. PMID 22939855
- [Derived] Pike NA, Pemberton V, Allen K, Jacobs JP, Hsu DT, Lewis AB, Ghanayem N, Lambert L, Crawford K, Atz T, Korsin R, Xu M, Ravishankar C, Cnota J, Pearson GD. Challenges and successes of recruitment in the "angiotensin-converting enzyme inhibition in infants with single ventricle trial" of the Pediatric Heart Network. Cardiol Young. 2013 Apr;23(2):248-57. doi: 10.1017/S1047951112000832. Epub 2012 Jul 5. PMID 22931751
- [Derived] Williams RV, Zak V, Ravishankar C, Altmann K, Anderson J, Atz AM, Dunbar-Masterson C, Ghanayem N, Lambert L, Lurito K, Medoff-Cooper B, Margossian R, Pemberton VL, Russell J, Stylianou M, Hsu D; Pediatric Heart Network Investigators. Factors affecting growth in infants with single ventricle physiology: a report from the Pediatric Heart Network Infant Single Ventricle Trial. J Pediatr. 2011 Dec;159(6):1017-22.e2. doi: 10.1016/j.jpeds.2011.05.051. Epub 2011 Jul 23. PMID 21784436
- [Derived] Mital S, Chung WK, Colan SD, Sleeper LA, Manlhiot C, Arrington CB, Cnota JF, Graham EM, Mitchell ME, Goldmuntz E, Li JS, Levine JC, Lee TM, Margossian R, Hsu DT; Pediatric Heart Network Investigators. Renin-angiotensin-aldosterone genotype influences ventricular remodeling in infants with single ventricle. Circulation. 2011 May 31;123(21):2353-62. doi: 10.1161/CIRCULATIONAHA.110.004341. Epub 2011 May 16. PMID 21576655
- [Derived] Hsu DT, Zak V, Mahony L, Sleeper LA, Atz AM, Levine JC, Barker PC, Ravishankar C, McCrindle BW, Williams RV, Altmann K, Ghanayem NS, Margossian R, Chung WK, Border WL, Pearson GD, Stylianou MP, Mital S; Pediatric Heart Network Investigators. Enalapril in infants with single ventricle: results of a multicenter randomized trial. Circulation. 2010 Jul 27;122(4):333-40. doi: 10.1161/CIRCULATIONAHA.109.927988. Epub 2010 Jul 12. PMID 20625111
- [Derived] Hsu DT, Mital S, Ravishankar C, Margossian R, Li JS, Sleeper LA, Williams RV, Levine JC, McCrindle BW, Atz AM, Servedio D, Mahony L; Pediatric Heart Network Investigators. Rationale and design of a trial of angiotensin-converting enzyme inhibition in infants with single ventricle. Am Heart J. 2009 Jan;157(1):37-45. doi: 10.1016/j.ahj.2008.08.030. PMID 19081394

RESULTS

PARTICIPANT FLOW:
Groups:
- Enalapril: ACE (Angiotensin-converting enzyme) inhibitor enalapril, initial dose 0.1 mg/kg/day; Uptitrated as tolerated to target dose of 0.4 mg/kg/day given in two divided doses
- Placebo: Placebo suspension
Period: Overall Study
Arm/Group | Enalapril | Placebo
Started | 115 | 115
Completed | 91 | 94
Not Completed | 24 | 21
Not completed — Death or Transplant | 14 | 16
Not completed — Family or MD withdrew subject | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enalapril | Placebo | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 115 | 115 | 230
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: days] | 20.1 (8.9) | 20.7 (9.1) | 20.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 28 | 68
  Male | 75 | 87 | 162
Race/Ethnicity, Customized [Number; unit: participants]
  White | 96 | 89 | 185
  Black/African-American | 12 | 20 | 32
  Asian | 4 | 3 | 7
  Other | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 104 | 105 | 209
  Canada | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Weight-for-age Z-score at 14 Months of Age
Description: Weight-for-age z-score at 14 months of age. In primary analysis outcome is defined as predicted mean of weight z-score at age 14 months based on longitudinal modeling(and adjusted for baseline values)
Time Frame: Measured at baseline, 2 weeks after starting study drug, just prior to the Glenn surgery, 7 days after restarting drug following the Glenn surgery, at 10 months of age, and at 14 months of age
Population: ITT, no imputation
Measure: Least Squares Mean (Standard Error); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 91 | 94
standard deviation | -0.62 (0.13) | -0.42 (0.13)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis; Mean Difference (Final Values) = -0.20, Standard Error of Mean 0.18

2. Secondary Outcome: Height-for-age Z-score
Description: Height-for-age z-score at 14 months of age. In primary analysis outcome is defined as predicted mean of height z-score at age 14 months based on longitudinal modeling (adjusted bor baseline value)
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 91 | 94
standard deviation | -1.00 (0.13) | -0.86 (0.13)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis; Mean Difference (Final Values) = -0.14

3. Secondary Outcome: Head Circumference-for-age Z-score
Description: Head circumference-for-age z-score at 14 months of age.In primary analysis outcome is defined as predicted mean of Head circumference z-score at age 14 months based on longitudinal modeling(and adjusted for baseline values)
Time Frame: as for outcome 1
Population: ITT, no imputation
Measure: Least Squares Mean (Standard Error); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 91 | 94
standard deviation | -0.55 (0.17) | 0.09 (0.17)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; Median Difference (Final Values) = -0.64

4. Secondary Outcome: Number of Participants With Ross Heart Failure Class I
Description: Class I is defined as having no limitations or symptoms of heart failure. Classes II to IV include increasing degrees of growth failure, prolonged feeding time, tachypnea, diaphoresis, and in older children, dyspnea on exercise.
Time Frame: Just prior to the pre-Glenn surgery
Population: Intention-to-treat analysis of participants measured just prior to the Glenn surgery
Measure: Number; unit: Participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 96 | 102
Participants | 53 | 56
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 1.00, Fisher Exact

5. Secondary Outcome: Number of Participants With Ross Heart Failure Class I
Description: as for outcome 4
Time Frame: Measured at 14 months of age
Population: Intention-to-treat analysis of participants completing the final study visit (target visit window age 14 months)
Measure: Number; unit: participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 91 | 94
participants | 72 | 77
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.71, Fisher Exact

6. Secondary Outcome: B-Type Natriuretic Peptide
Description: B-Type Natriuretic Peptide (BNP) level.
Time Frame: Measured just prior to the Glenn surgery
Population: ITT analysis, no imputation
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 83 | 90
pg/ml | 79 [30 to 182] | 84 [36 to 196]
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.74, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: B-type Natriuretic Peptide Level
Description: B-type natriuretic peptide (BNP) level.
Time Frame: at the time of the 14 month visit
Population: ITT, no imputation
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 69 | 65
pg/ml | 25 [13 to 35] | 39 [21 to 86]
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.22, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Neurodevelopmental Status (PDI): the Bayley Scales of Infant Development,Psychomotor Development Index Z-score
Description: Neurodevelopmental status (PDI):
  the Bayley Scales of Infant Development: Psychomotor Development index z-score .
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 86 | 83
standard deviation | -1.29 (1.19) | -1.32 (1.22)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.86, t-test, 2 sided

9. Secondary Outcome: Neurodevelopmental Status(MDI): Bayley Scales of Infant Development, Mental Developmental Index Z-score
Description: Neurodevelopmental status(MDI):Bayley Scales of infant development, Mental Developmental Index z-score .
Time Frame: at 14 months of age
Population: ITT, not imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 83
standard deviation | -0.26 (0.91) | -0.33 (1.02)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.60, t-test, 2 sided

10. Secondary Outcome: Neurodevelopmental Status (FSII)
Description: Functional status II (Revised) Total Score. Scale ranges up to 100.00, the higher the better. The score presents an instrument for assessing health status for children surviving long term with chronic physcial disorders.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 89 | 89
units on a scale | 96.4 [89 to 100] | 96.4 [86 to 100]
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.60, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: MacArthur-Bates Inventory -Phrases Understood
Description: MacArthur-Bates Communicative Development inventory( Words and Gestures)-Phrases Understood z-score.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 90 | 87
standard deviation | -0.48 (1.11) | -0.92 (1.17)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.01, t-test, 2 sided

12. Secondary Outcome: MacArthur-Bates Inventory -Words Understood
Description: MacArthur-Bates Communicative Development inventory( Words and Gestures)-Words Understood z-score.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 90 | 87
standard deviation | -0.46 (0.91) | -0.82 (0.83)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.008, t-test, 2 sided

13. Secondary Outcome: MacArthur-Bates Inventory -Total Gestures
Description: MacArthur-Bates Communicative Development inventory( Words and Gestures)-Total Gestures z-score.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 90 | 87
standard deviation | -0.86 (1.07) | -1.31 (0.97)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

14. Secondary Outcome: MacArthur-Bates Inventory -Words Produced
Description: MacArthur-Bates Communicative Development inventory( Words and Gestures)-Words Produced z-score.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Median (Inter-Quartile Range); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 90 | 87
standard deviation | -0.60 [-0.72 to 0.41] | -0.63 [-0.75 to 0.42]
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.31, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Ejection Fraction (%)
Description: Two-dimensional echocardiography endpoint -Total Ejection Fraction (%) per Core Laboratory assessment. Ejection Fraction % is defined as the percentage of the stroke volume (i.e. difference between end-diastolic and end-systolic volumes) in a ventricle relative to end-diastolic volume.
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: percent (of end diastolic volume)
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 94 | 95
percent (of end diastolic volume) | 57.9 (9.8) | 56.6 (10.2)
Statistical Analysis 1: Comparison: Enalapril; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

16. Secondary Outcome: Ejection Fraction (%)
Description: Two-dimensional echocardiography endpoint -Total Ejection Fraction (%) per Core Laboratory assessment. Ejection Fraction (%) is defined as percentage of stroke volume of a ventricle (i.e. the difference between end diastolic and end systolic volumes)relative to end diastolic volume.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: percent (of end diastolic volume)
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 91
percent (of end diastolic volume) | 59.3 (9.6) | 57.9 (10.4)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.37, t-test, 2 sided

17. Secondary Outcome: Ventricular Mass
Description: Two-dimensional echocardiography endpoint - Total Ventricular mass (g) per Core Laboratory assessment.
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 93 | 94
g | 25.5 (9.2) | 28.1 (10.6)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.08, t-test, 2 sided

18. Secondary Outcome: Ventricular Mass
Description: Two-Dimensional Echocardiography endpoint-Total Ventricular mass (g) per Core Laboratory assessment. Range from 15.60 to 70.40
Time Frame: At 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 89
g | 31.4 (10.3) | 34.4 (11.4)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.07, t-test, 2 sided

19. Secondary Outcome: Ventricular Mass Z-score
Description: Two-dimensional echocardiography endpoint -Total Ventricular mass z-score per Core Laboratory assessment.
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 92 | 92
standard deviation | 4.0 (2.9) | 4.9 (3.3)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

20. Secondary Outcome: Ventricular Mass Z-score
Description: Two-dimensional echocardiography endpoint -Total Ventricular mass z-score per Core Laboratory assessment.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 89
standard deviation | 2.5 (2.3) | 3.1 (2.5)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

21. Secondary Outcome: End-diastolic Volume
Description: Two-Dimensional Echocardiography endpoint - Total End-diastolic volume (ml) per Core Laboratory assessment.
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 94 | 95
ml | 24.1 (10.1) | 23.2 (9.0)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.49, t-test, 2 sided

22. Secondary Outcome: End-diastolic Volume
Description: Two-Dimensional Echocardiography endpoint - Total End-diastolic volume (ml) per Core Laboratory assessment.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 91
ml | 29.2 (10.0) | 30.7 (11.3)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.35, t-test, 2 sided

23. Secondary Outcome: End Diastolic Volume Z-score
Description: Two-dimensional echocardiography endpoint -total End diastolic volume z-score per Core Laboratory assessment.
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 93 | 93
standard deviation | 2.3 (2.5) | 2.1 (2.5)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.62, t-test, 2 sided

24. Secondary Outcome: End-diastolic Volume Z-score
Description: Two-dimensional echocardiography endpoint -total end-diastolic volume z-score per Core Laboratory assessment.
Time Frame: at 14 months of age
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: standard deviation
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 91
standard deviation | 1.1 (2.1) | 1.3 (2.4)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.43, t-test, 2 sided

25. Secondary Outcome: Ventricular Mass to Volume Ratio
Description: Two-Dimensional Echocardiography endpoint -Ventricular Mass to Volume ratio per Core Laboratory assessment.
Time Frame: Measured just before the Glenn surgery
Population: Intention-to-treat analysis of participants completing the pre-Glenn visit
Measure: Mean (Standard Deviation); unit: g/ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 93 | 94
g/ml | 1.15 (0.43) | 1.31 (0.50)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.02, t-test, 2 sided

26. Secondary Outcome: Ventricular Mass to Volume Ratio
Description: Two-Dimensional Echocardiography endpoint -Ventricular Mass to Volume ratio per Core Laboratory assessment.
Time Frame: Measured at 14 months of age
Population: Intention-to-treat analysis of participants completing the final study visit (target visit window age 14 months)
Measure: Mean (Standard Deviation); unit: g/ml
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 87 | 89
g/ml | 1.14 (0.38) | 1.20 (0.44)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.34, t-test, 2 sided

27. Secondary Outcome: Ventricular Filling Pressure
Description: Ventricular filling pressure measured by catherization
Time Frame: just before the Glenn surgery
Population: ITT, no imputation
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 58 | 63
mmHg | 10.9 (3.6) | 11.1 (4.0)
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = .81, t-test, 2 sided

28. Secondary Outcome: Number of Participants With Moderate to Severe AV Valve Regurgitation
Description: Number of participants with Moderate to severe AV valve regurgitation.
Time Frame: just before the pre-Glenn surgery
Population: ITT, no imputation
Measure: Number; unit: participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 98 | 98
participants | 20 | 32
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.08, Fisher Exact

29. Secondary Outcome: Number of Participants With Moderate to Severe AV Valve Regurgitation
Description: Number of participants with moderate to severe AV valve regurgitation.
Time Frame: at age 14 months
Population: ITT, no imputation
Measure: Number; unit: participants
Arm/Group | Enalapril | Placebo
Number analyzed (Participants) | 90 | 93
participants | 11 | 22
Statistical Analysis 1: Comparison: Enalapril vs Placebo; Test type: Superiority or Other; p = 0.06, Fisher Exact

ADVERSE EVENTS:
Time Frame: Randomization to 14 months of age
Description: All serious AE counts by body system are presented. The total count of affected by SAE is based on all reported SAEs.
  All other AE counts by body system are presented. The total count of affected by "other AE" is based on all reported AEs other than serious.
Arm/Group | Enalapril | Placebo
Serious Adverse Events (participants affected / at risk) | 88/115 | 87/115
Other Adverse Events (participants affected / at risk) | 77/115 | 70/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enalapril (N=115) | Placebo (N=115)
Cardiac general (Cardiac disorders) | 29 (37) | 19 (24) — Adjudication by independent medical monitor for all serious adverse events
Infection (Infections and infestations) | 36 (55) | 35 (44)
Neurology (Nervous system disorders) | 4 (4) | 6 (6)
Pulmonary/Upper Respiratory (Respiratory, thoracic and mediastinal disorders) | 31 (41) | 35 (49)
Vascular (Vascular disorders) | 22 (30) | 21 (26)
auditory/ear (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Adjudication by independent medical monitor for all serious adverse events
blood/bone marrow (Blood and lymphatic system disorders) | 4 (4) | 2 (2) — Adjudication by independent medical monitor for all serious adverse events
cardiac arrhythmia (Cardiac disorders) | 4 (5) | 5 (6) — Adjudication by independent medical monitor for all serious adverse events
coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Adjudication by independent medical monitor for all serious adverse events
constitutional symptoms (General disorders) | 2 (2) | 3 (3) — Adjudication by independent medical monitor for all serious adverse events
death (Cardiac disorders) | 5 (5) | 4 (4) — Adjudication by independent medical monitor for all serious adverse events
dermatology/skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Adjudication by independent medical monitor for all serious adverse events
gastrointestinal (Gastrointestinal disorders) | 20 (27) | 18 (26) — Adjudication by independent medical monitor for all serious adverse events
growth and development (Metabolism and nutrition disorders) | 1 (1) | 5 (5) — Adjudication by independent medical monitor for all serious adverse events
hemorrhage/bleeding (Blood and lymphatic system disorders) | 1 (1) | 2 (2) — Adjudication by independent medical monitor for all serious adverse events
lymphatics (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Adjudication by independent medical monitor for all serious adverse events
metabolic/laboratory (Metabolism and nutrition disorders) | 3 (3) | 0 (0) — Adjudication by independent medical monitor for all serious adverse events
musculoskeletal/soft issue (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) — Adjudication by independent medical monitor for all serious adverse events
renal/genitourinary (Renal and urinary disorders) | 1 (1) | 1 (2) — Adjudication by independent medical monitor for all serious adverse events
surgery/intra-operative injury (Surgical and medical procedures) | 0 (0) | 3 (3) — Adjudication by independent medical monitor for all serious adverse events
syndromes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Adjudication by independent medical monitor for all serious adverse events
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enalapril (N=115) | Placebo (N=115)
Cardiac General (Cardiac disorders) | 18 (23) | 12 (15)
Neurology (Nervous system disorders) | 5 (6) | 6 (9)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 22 (25)
Vascular (Vascular disorders) | 7 (7) | 5 (5)
infection (Infections and infestations) | 38 (66) | 33 (64)
allergy/immunology (Immune system disorders) | 1 (1) | 2 (3)
auditory/ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
blood/bone marrow (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
cardiac arrhythmia (Cardiac disorders) | 10 (12) | 5 (6)
coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
constitutional symptoms (General disorders) | 8 (8) | 3 (4)
dermatology/skin (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (9)
endocrine (Endocrine disorders) | 2 (2) | 0 (0)
gastrointestinal (Gastrointestinal disorders) | 19 (27) | 16 (24)
hemorrhage/bleeding (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
hepatobillary (Hepatobiliary disorders) | 2 (2) | 0 (0)
metabolic/laboratory (Metabolism and nutrition disorders) | 7 (8) | 9 (9)
renal/genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
surgery/intra-operative injury (Surgical and medical procedures) | 2 (2) | 0 (0)
growth and development (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
musculoskeletal/soft tissue (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No